CLINICAL TRIAL: NCT02650011
Title: The Clinical Features and Natural History of Acute-on-Chronic Liver Failure in Korean Patients With Chronic Liver Disease: Multicenter, Prospective Cohort Study
Brief Title: Clinical Features and Natural History of Acute-on-Chronic Liver Failure in Korean Patients With Chronic Liver Disease
Status: Suspended | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Dong Joon Kim, Professor and Chief, Division of Gastroenterology and Hepatology Hallym University College of Medicine / Director, Center for Liver and Digestive Diseases Hallym University Medical Center, Chuncheon Sacred Heart Hospital
Other Study IDs: P-KACLiF
Record Dates: First submitted 2015-07-25; First posted 2016-01-08 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Chronic Liver Disease; Acute Derangement of Liver Function
Keywords: Chronic liver disease; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACLF cohort: Patients who have chronic liver disease and admitted for acute deterioration of liver function
  Interventions: Other: Acute deterioration of liver function

INTERVENTIONS:
Other: Acute deterioration of liver function — development of new ascites within 4 weeks or re-emergence of ascites who have previous well controlled ascites (greater than or equal to grade 2 or 3; International ascites club criteria) development of hepatic encephalopathy development of gastrointestinal hemorrhage development of jaundice (serum bilirubin greater than or equal to 3mg/dl) development of bacterial infection

SUMMARY:
Chronic liver disease including liver cirrhosis is still associated with high mortality, although advancement of medical management and transplantation. Acute-on-chronic liver failure (ACLF) refers to condition of previously stable chronic liver disease with occurrence of an acute insult resulting in rapid deterioration of liver function and subsequent decompensation. This condition is different from liver cirrhosis (chronic hepatic decompensation) in terms of having more chance of recovery with management before acute deterioration, although it shows high short-term mortality. Thus, earlier recognition and intensive management are important for this condition. However, the definition or diagnostic criteria is unclear and the natural course of this condition is not definitely investigated. The aim of this study is to establish the natural course of ACLF in Korean patients.

DETAILED DESCRIPTION:
Chronic liver disease including liver cirrhosis is still associated with high mortality, although advancement of medical management and transplantation. Acute-on-chronic liver failure (ACLF) refers to condition of previously stable chronic liver disease with occurrence of an acute insult resulting in rapid deterioration of liver function and subsequent decompensation. Various factors could be a precipitating factor of ACLF. This condition is different from liver cirrhosis (chronic hepatic decompensation) in terms of having more chance of recovery with management before acute deterioration, although it shows high short-term mortality. Thus, earlier recognition and intensive management are important for this condition. However, the definition or diagnostic criteria is unclear and the natural course of this condition is not definitely investigated. The aim of this study is to establish the common etiology, symptom and natural course of ACLF in Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease: Chronic hepatitis B, Chronic hepatitis C, Alcoholic liver disease, Biopsy proven or clinically diagnosed liver cirrhosis, Other chronic liver diseases including non-alcoholic fatty liver disease, primary biliary cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, a-1 antitrypsin deficiency, and cryptogenic causes.
* Acute deterioration of liver function: more than one of the below criteria

  1. development of new ascites within 4 weeks or re-emergence of ascites who have previous well controlled ascites (greater than or equal to grade 2 or 3; International ascites club criteria)
  2. development of hepatic encephalopathy
  3. development of gastrointestinal hemorrhage
  4. development of jaundice (serum bilirubin greater than or equal to 3mg/dl)
  5. development of bacterial infection
* spontaneous bacteremia: positive blood cultures without a source of infection
* spontaneous bacterial peritonitis: ascitic fluid polymorphonuclear cells >250/µL
* lower respiratory tract infections: new pulmonary infiltrate in the presence of: i) at least one respiratory symptom (cough, sputum production, dyspnea, pleuritic pain) with ii) at least one finding on auscultation (rales or crepitation) or one sign of infection (core body temperature >38_C or less than 36_C, shivering, or leukocyte count >10,000/mm3 or <4,000/mm3) in the absence of antibiotics
* Clostridium difficile Infection: diarrhea with a positive C. difficile assay
* bacterial entero-colitis: diarrhea or dysentery with a positive stool culture for Salmonella, Shigella, Yersinia, Campylobacter, or pathogenic E. coli;
* soft-tissue/skin Infection: fever with cellulitis
* urinary tract infection (UTI): urine white blood cell >15/high-power field with either positive urine gram stain or culture;
* intra-abdominal infections: diverticulitis, appendicitis, cholangitis, etc.
* other infections not covered above;
* fungal infections as a separate category.

Exclusion Criteria:

* Patients who do not have chronic liver disease
* Patients who have hepatocellular carcinoma
* Patients who admitted for extrahepatic manifestations
* Patients who have HIV infection
* Patients who admitted for symptomatic control of chronic liver disease, other than acute deterioration of liver function

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have chronic liver disease and admitted for acute deterioration of liver function (ACLF)
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall mortality of patients with ACLF | up to 21 months
  Overall mortality of ACLF in original cohort

SECONDARY OUTCOMES:
Overall rate of liver transplantation in patients with ACLF | up to 21 months
  Overall rate of liver transplantation in original cohort
Short term mortality of patients with ACLF | 28 day and 90 day of observation
  Short term mortality of ACLF in original cohort
Short term rate of liver transplantation in patients with ACLF | 28 day and 90 day of observation
  Short term rate of liver transplantation in original cohort

CONTACTS AND LOCATIONS:
Overall Officials: Dong Joon Kim, M.D., Ph.D., Principal Investigator — Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, South Korea

REFERENCES:
- [Derived] Kim TH, Yim HJ, Jung YK, Song DS, Yoon EL, Kim HY, Kang SH, Chang Y, Yoo JJ, Jun BG, Lee SW, Park JG, Park JW, Kim SE, Kim TY, Jeong SW, Suk KT, Kim MY, Kim SG, Kim W, Jang JY, Yang JM, Kim DJ; Korean Acute-on-Chronic Liver Failure (KACLiF) Study Group. New prognostic model for hospitalized patients with alcoholic cirrhosis and Maddrey's discriminant function <32. Hepatol Int. 2024 Apr;18(2):500-508. doi: 10.1007/s12072-023-10582-1. Epub 2023 Oct 13. PMID 37831433